CLINICAL TRIAL: NCT03966404
Title: EyeBOX Concussion Study and Registry
Status: Completed | Type: Observational
Sponsor: Oculogica, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: MTBI002
Record Dates: First submitted 2019-05-22; First posted 2019-05-29 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Concussion, Brain; Mild Traumatic Brain Injury
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

INTERVENTIONS:
Diagnostic Test: EyeBOX device — The EyeBOX medical device tracks a patient's eye movement and calculates a BOX Score ranging from 0-20. The BOX score is interpreted as a binary classification for eye movement abnormalities, where anything equal to or greater than 10 is a positive result for the initial evaluation of concussion and everything below 10 is negative.

SUMMARY:
The objective of this study is to further evaluate eye movements as an aid in the diagnosis of concussion / mTBI and the utility of eye movement assessment in the monitoring of symptoms over time after an initial diagnosis of concussion.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent or assent along with guardian consent.
2. Have sustained a suspected direct or indirect force to the head with or without documented loss of consciousness, memory loss, alteration in consciousness or neurologic deficits. Only individuals presenting for initial evaluation of concussion may be enrolled, however longitudinal assessments may be conducted on enrolled subjects.
3. Have the ability to provide a complete ophthalmologic, medical and neurologic history as well as report medications/drugs/alcohol consumed within the 24 hours prior to tracking.

Exclusion Criteria:

1. Have penetrating trauma.
2. Have had a conventional head CT or MRI demonstrating evidence of structural brain injury (subdural, epidural or intraparenchymal hemorrhage, edema/mass effect per attending radiologist read).
3. Either of the following conditions, immediately related to the incident head trauma: loss of consciousness exceeding 30 minutes or best available GCS score less than 13 within 24 hours.
4. Be blind (no light perception), have missing or non-functional eyes.
5. Be unable to open their eyes.
6. Have a history of unresolved strabismus, diplopia, amblyopia.
7. Have a history of unresolved cranial nerve III, IV, or VI palsy.
8. Have a history of unresolved macular edema, retinal degeneration, extensive cataract, or ocular globe disruption.
9. Have a history of extensive prior eye surgery (examples include strabismus surgery, scleral buckle repair of retinal detachment, repair of blow out fractures of the orbit and any procedures that would interfere with extraocular muscle movements; prior cataract surgery or Lasik are not exclusions) or scarring.
10. Have a prior history of unresolved ocular-motor dysfunctions.
11. Be intoxicated.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: All consecutive subjects who meet all of the inclusion criteria and none of the exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2019-08-05 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
diagnostic accuracy of initial clinical diagnosis of concussion | day 0 (when patient first presents for evaluation)
  sensitivity and specificity compared to initial clinical diagnosis of concussion
diagnostic accuracy of clinical diagnosis of post-concussion symptoms | up to one year after initial presentation
  sensitivity and specificity compared to clinical diagnosis of post-concussion symptoms
adverse events | through study participation, up to one year
  adverse events occurring during use of the diagnostic device

SECONDARY OUTCOMES:
diagnostic accuracy of initial clinical diagnosis of concussion | day 0 (when patient first presents for evaluation)
  positive and negative predictive value compared to initial clinical diagnosis of concussion
correlation with increases or decreases in post-concussion symptom severity | up to one year after initial presentation
  diagnostic accuracy to identify increases or decreases in post-concussion symptom severity

CONTACTS AND LOCATIONS:
Overall Officials: Rosina Samadani, PhD, Study Director — Oculogica, Inc.
Locations (1):
- New York Sports Medicine Institute, White Plains, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided